CLINICAL TRIAL: NCT05803525
Title: كفاءة الدعامات و هيبوكلوريت الصوديوم مجتمعة في التجديد اللبى للأسنان الغير مكتملة
Brief Title: Efficacy of Combined Scaffolds and Sodium Hypochlorite in Regenerative Endodontics of Immature Teeth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Hanan Mohamed Arb, Assistant professor in Endodontic department Tanta University, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HananArb
Record Dates: First submitted 2022-12-10; First posted 2023-04-07 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-03

CONDITIONS: Incomplete Root Formation of Anterior Teeth

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Double (Investigator, Outcomes Assessor)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- • Group I: BC scaffold and 0.5% concentration of NaOCl irrigant solution. (Active Comparator): BC will be made & use 0.5 NaOCl conc
  Interventions: Other: Intra-canal medication protocol
- • Group II: BC scaffold and 2.5% concentration of NaOCl irrigant solution. • (Active Comparator): BC will be made & use 2.5 NaOCl conc
  Interventions: Other: Intra-canal medication protocol
- • Group III: PRF scaffold and 0.5% concentration of NaOCl irrigant solution. • (Active Comparator): PRF will be made & use 0.5 NaOCl conc
  Interventions: Other: Intra-canal medication protocol
- Group IV: PRF scaffold and 2.5% concentration of NaOCl irrigant solution. • (Active Comparator): PRF will be made & use 2.5 NaOCl conc
  Interventions: Other: Intra-canal medication protocol
- • Group V: Collagen scaffold and 0.5% concentration of NaOCl irrigant solution. (Active Comparator): Collagen will be made & use 0.5 NaOCl conc
  Interventions: Other: Intra-canal medication protocol
- • Group VI: Collagen scaffold and 2.5% concentration of NaOCl irrigant solution. (Active Comparator): Collagen will be made & use 2.5 NaOCl conc
  Interventions: Other: Intra-canal medication protocol

INTERVENTIONS:
Other: Intra-canal medication protocol — Copious gentle irrigation will be provided without canal instrumentation using 20 mL 1.5% NaOCl in a slow flowing rate by a 27-gauge irrigating side vented needle positioned 2 mm from the root end followed by 20 mL saline.
  After root canal dryness using paper points , double antibiotic paste (DAP) containing 500 mg of metronidazole and ciprofloxacin mixed with 0.5 mL polypropylene glycol giving a creamy paste will transported into root canal via lentulo spiral filler positioned 2 mm shorter than the WL apically and to level just below the cement-enamel junction (CEJ) coronally. Access cavity will be sealed response to the initial treatment will be assessed after 3 weeks.(21) In the next visit, If the patient is asymptomatic, the DAP will be removed using 10 mL of NaOCl according to the concentrations mentioned in each study group, followed by copious irrigation with 10 mL of 17% EDTA (22) and normal saline then drying the canals with sterile paper points.

SUMMARY:
The aim of the study is to evaluate the efficacy of combinations of different scaffolds (blood clot, platelet rich fibrin, collagen) and sodium hypochlorite concentrations (0.5%- 2.5%) in regenerative endodontics of immature non-vital anterior teeth clinically and radiographically using cone-beam computed tomography.

DETAILED DESCRIPTION:
Patients will be divided randomly into six equal groups (n=8)

* Group I: BC scaffold and 0.5% concentration of NaOCl irrigant solution.
* Group II: BC scaffold and 2.5% concentration of NaOCl irrigant solution.
* Group III: PRF scaffold and 0.5% concentration of NaOCl irrigant solution.
* Group IV: PRF scaffold and 2.5% concentration of NaOCl irrigant solution.
* Group V: Collagen scaffold and 0.5% concentration of NaOCl irrigant solution.
* Group VI: Collagen scaffold and 2.5% concentration of NaOCl irrigant solution.

CBCT image will be obtained for baseline records after placement of the final resin restoration then the patients will be recalled after 6 months and 12 months for evaluating any changes in root length, root canal width, apex diameter and lesion size if present. The success rates for patients at each recall visit will be scored as follows

1. Score 0: Persistence of clinical and radiographic findings.
2. Score 1: Absence of swelling, drainage and pain along with radiographic evidence of osseous healing + no evidence of increased root dimensions.
3. Score 2: Absence of swelling, drainage and pain along with radiographic evidence of osseous healing + radiographic root development.

ELIGIBILITY:
Inclusion Criteria:

* • Patients, abarantly free from any systemic diseases that may hinder the normal healing process.

  * Maxillary traumatized or cariously exposed immature anterior teeth.
  * Clinical signs of pulp necrosis.
  * Radiographic evidence of incomplete root development based on an apical opening >1 mm.

Exclusion Criteria:

* • Allergy to medication used in the procedure or any medical conditions that contraindicate endodontic treatment (eg, acute systemic disease and abnormalities in host defense).

  * Non-restorable tooth.
  * Radiographic evidence of root fracture.
  * Lack of patient and parent cooperation.
  * Teeth with vital pulps and complete root development.
  * Presence of periodontal pocket > 4 mm.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2020-01-15 (Actual); Primary Completion 2023-08-15 (Estimated); Study Completion 2024-01-30 (Estimated)

PRIMARY OUTCOMES:
diameter of periapical radiolucency | 1 year
  radiographic changes in root
diameter of root length | 1 year
  radiographic changes in root

SECONDARY OUTCOMES:
Pain scale | 1 year
visual changes in discoloration | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Tanta University, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No